CLINICAL TRIAL: NCT03197558
Title: A Prospective, Multicenter Study to Evaluate Effectiveness and Safety of Lidocaine Iontophoresis and Tympanostomy Tube Placement Using the Tula Iontophoresis and Tube Delivery Systems for Adults in an Office Setting
Brief Title: Adult Study to Evaluate Placement of Tympanostomy Tubes In-office (ADEPT)
Acronym: ADEPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tusker Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR007003 - Group B
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Barotrauma;Ear; OME - Otitis Media With Effusion; AOM - Acute Otitis Media; Eustachian Tube Dysfunction
MeSH Terms: conditions — Otitis Media with Effusion; Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Tube insertion using Tube Delivery System (TDS) (Other): Active Tymbion iontophoresis and tube insertion using the TDS
  Interventions: Combination Product: Tymbion Iontophoresis and Tube Delivery System (TDS)

INTERVENTIONS:
Combination Product: Tymbion Iontophoresis and Tube Delivery System (TDS) — Subjects will receive active Tymbion iontophoresis and tube insertion using the Tube Delivery System in all ears indicated for tube placement.

SUMMARY:
A prospective, multicenter study to evaluate effectiveness and safety of Tymbion iontophoresis and tympanostomy tube placement using the Tula iontophoresis and tube delivery systems for adults in an office setting.

This study cohort is called Group B and includes tube placement. Protocol CPR007003 also included a first study group ('A', without tube placement) that was completed and described in a separate registration (NCT03119181).

DETAILED DESCRIPTION:
The objective for Group B in the study is to evaluate tolerability and safety of tympanostomy tube (TT) placement in adults following local anesthesia in a physician's clinic setting.

Group B will consist of 30 evaluable adults who require unilateral or bilateral tube insertion.

The iontophoresis system (IPS) will be used to facilitate anesthetic delivery to the tympanic membrane (TM). The lidocaine-based solution used for local anesthesia of the TM is Tymbion (2% lidocaine HCl/ 1:100,000 epinephrine).

Subjects will receive active Tymbion iontophoresis and will have tubes placed using the TDS in all ears indicated for tube placement. The subject will rate the pain upon TDS tube insertion using the VAS, and the pain score will be compared to a performance goal.

Safety will be evaluated post procedure and at a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 18 years of age at time of consent
2. Indication for tympanostomy tube insertion per Clinical Practice Guideline,or indicated for tympanostomy tube insertion due to barotrauma or Eustachian tube dysfunction per AAO-HNS Clinical Indicators.
3. Subject is able and willing to comply with the protocol and attend all study visits.
4. Subject is able and willing to provide informed consent.
5. Subject is able to read and understand English.

Exclusion Criteria by Ear:

1. Significantly atrophic, retracted or retraction pocket at location of tube placement, bimeric, monomeric or atelectatic tympanic membrane.
2. Perforated tympanic membrane.
3. Otitis externa.
4. Hemotympanum.
5. Damaged/denuded skin in the auditory canal.
6. Cerumen impaction resulting in a significant amount of cleaning required to visualize the tympanic membrane potentially causing abrasion or irritation to the external ear canal.
7. Notable ear discomfort experienced during audiologic or otoscopic examination.
8. Anatomy that precludes sufficient visualization of and access to the tympanic membrane.
9. Anatomy that necessitates tympanostomy tube placement in the posterior half of the tympanic membrane.

   General Exclusion Criteria
10. Pregnant or lactating females
11. History of sensitivity or allergic reaction to lidocaine HCl, tetracaine, epinephrine, or any hypersensitivity to local anesthetics.
12. Familial history of insensitivity to lidocaine or other local anesthetics of the amide type.
13. Electrically sensitive medical support systems (eg, pacemakers, defibrillators, cochlear implants)
14. Other conditions that would preclude performing the study procedure including iontophoresis system ear plug incompatibility.
15. Health conditions that, in the opinion of the investigator, would present undue risk to the subject, based on device/anesthetic drug product label warnings and precautions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Yen, MD, Principal Investigator — Specialty Physician Associates
Locations (8):
- United States (8):
  - Sacramento ENT, Roseville, California
  - Camino ENT, San Jose, California
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Charlotte Eye Ear Nose and Throat Associates, Charlotte, North Carolina
  - Specialty Physician Associates, Bethlehem, Pennsylvania
  - South Carolina ENT, Lugoff, South Carolina
  - Carolina Ear, Nose and Throat, Orangeburg, South Carolina
  - Ear Medical Group, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tube Insertion Using Tube Delivery System (TDS): Active Tymbion iontophoresis and tubes using the TDS
  Tymbion Iontophoresis and Tube Delivery System (TDS): Subjects will receive active Tymbion iontophoresis and will have tubes placed using the TDS in all ears indicated for tube placement.
Period: Overall Study
Arm/Group | Tube Insertion Using Tube Delivery System (TDS)
Started | 30
Completed (Participants undergoing iontophoresis with adequate anesthesia for tube placement.) | 29
Not Completed | 1
Not completed — Tubes not placed | 1

BASELINE CHARACTERISTICS:
Population: Participants for whom iontophoresis is initiated.
Arm/Group | Tube Insertion Using Tube Delivery System (TDS)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 21
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Subject-reported Pain Score Following Tube Delivery System (TDS) Tube Placement Using the Visual Analogue Scale (VAS) by Subject Compared to a Performance Goal.
Description: The VAS consists of a 100 millimeter (mm) line with a statement at each end representing the extreme limits of pain intensity where a score of 0 represents "No pain" and a score of 100 represents "The worst possible pain".
  Following TDS tube placement, the subject will report their post-tube placement ear discomfort for each ear undergoing tube placement using the VAS. For subjects treated bilaterally, the highest (worst) score reported will be used as the unit of analysis.
Time Frame: Day of procedure (Day 0)- Immediately after tube placement
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Tube Insertion Using Tube Delivery System (TDS)
Number analyzed (Participants) | 29
millimeters | 9.4 (15.7)
Statistical Analysis 1: Comparison: Tube Insertion Using Tube Delivery System (TDS); Mean VAS score compared to performance goal using a bootstrap method test at 2.5% significance; Test type: Superiority — Upper confidence limit of mean VAS score hypothesized to be less than (superior) to a performance goal of 45 mm; Bootstrap method = 14.35, 97.5% CI 1-sided [upper limit 14.35]

ADVERSE EVENTS:
Time Frame: Procedure through 3-week post-procedure follow-up visit.
Arm/Group | Tube Insertion Using Tube Delivery System (TDS)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 10/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tube Insertion Using Tube Delivery System (TDS) (N=30)
Inadequate anesthesia (Ear and labyrinth disorders) | 1 (1) — Potentially related to procedure, device or drug
Ear discomfort (Ear and labyrinth disorders) | 1 (1) — Potentially related to procedure, device or drug
Tube in middle ear (Ear and labyrinth disorders) | 1 (1) — Potentially related to procedure, device or drug
Vertigo (Ear and labyrinth disorders) | 1 (1) — Potentially related to procedure, device or drug
Dizziness (Ear and labyrinth disorders) | 1 (1) — Potentially related to procedure, device or drug
Tube occlusion (Ear and labyrinth disorders) | 2 (2) — Potentially related to procedure, device or drug
Dehydration (Metabolism and nutrition disorders) | 1 (1) — Not related to procedure, device or drug
Otorrhea (Ear and labyrinth disorders) | 1 (1) — Not related to procedure, device or drug
Incontinence (Renal and urinary disorders) | 1 (1) — Not related to procedure, device or drug
Change in respiration rate (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Not related to procedure, device or drug. Per protocol, required to report any change in respiration > 30% as an adverse event. These events were not clinically significant and within normal range.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must submit communications to Sponsor for review and comment to verify accurate content at least 30 days prior to submitting to any third party. A delay up to 90 days may be requested by Sponsor in order to file patent applications relating to an Invention if applicable. Sponsor and PI agree that any Institution Publication shall only be made after the Multicenter Publication, provided that the Multicenter Publication is submitted within 18 months after conclusion of the study at all sites.

DOCUMENTS (2):
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT03197558/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT03197558/SAP_001.pdf